CLINICAL TRIAL: NCT03169101
Title: Understanding the Role of Cognitive Dysfunction in the Treatment of Nicotine Dependence Among HIV-infected Smokers
Brief Title: Cognition and Smoking Relapse (HCS)
Acronym: HCS
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 824860; R01DA042682 (NIH)
Record Dates: First submitted 2017-05-02; First posted 2017-05-30 (Actual); Results first posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-04

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; HIV; Cognition
MeSH Terms: conditions — Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine; Behavior Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two samples (one 10 mL and one 8 mL) of blood will be drawn at the Intake visit to evaluate the nicotine metabolite ratio and neuroinflammatory markers. All specimens are to be collected solely for research purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- HIV+ Smoking lab session first: HIV-infected smokers: diagnosed with HIV infection and exhibiting viral load of less than or equal to 1000 copies/mL and CD4+ counts of greater than or equal to 200 cells/mm3 within 6 months prior to enrollment Randomized to complete smoking-as-usual lab session first and 24-h abstinent lab session second
  Interventions: Drug: Nicotine patch; Behavioral: Behavioral counseling
- HIV- Smoking lab session first: HIV-uninfected smokers: negative HIV status will be confirmed by an on-site rapid HIV blood test Randomized to complete smoking-as-usual lab session first and 24-h abstinent lab session second
  Interventions: Drug: Nicotine patch; Behavioral: Behavioral counseling
- HIV+ Abstinent lab session first: HIV-infected smokers: diagnosed with HIV infection and exhibiting viral load of less than or equal to 1000 copies/mL and CD4+ counts of greater than or equal to 200 cells/mm3 within 6 months prior to enrollment Randomized to complete 24-h abstinent lab session first and smoking-as-usual lab session second
  Interventions: Drug: Nicotine patch; Behavioral: Behavioral counseling
- HIV- Abstinent lab session first: HIV-uninfected smokers: negative HIV status will be confirmed by an on-site rapid HIV blood test Randomized to complete 24-h abstinent lab session first and smoking-as-usual lab session second
  Interventions: Drug: Nicotine patch; Behavioral: Behavioral counseling

INTERVENTIONS:
Drug: Nicotine patch — All participants will receive nicotine patches to aid in quitting smoking. TN is available over the counter and is very well tolerated. Participants will use "the patch" in a tapering fashion as recommended by the manufacturer. Participants who smoke 10 or more cigarettes per day will adhere to the following dosing guidelines: 21 mg for 4 weeks; 14 mg for 2 weeks and 7 mg for 2 weeks. Individuals who smoke between 5 and 9 cigarettes per day will follow a modified dosing regimen: 14 mg for 6 weeks and 7 mg for 2 weeks.
  Other Names: Nicoderm CQ
Behavioral: Behavioral counseling — Participants will attend 6 counseling sessions and receive standard smoking cessation counseling (SC).

SUMMARY:
This study tests whether withdrawal-related cognitive deficits increase smoking relapse among HIV-infected (HIV+) vs. HIV-uninfected smokers (HIV-). Adult smokers (N=300; 150 HIV+, 150 HIV-) will complete 2 sessions to assess cognition (24h abstinence vs. smoking-as-usual; order counterbalanced; weeks 0-2). Subjects will then receive smoking cessation counseling and open label transdermal nicotine (weeks 3-12). Outcomes are: 1) cognition; and 2) abstinence rates at the end-of-treatment.

DETAILED DESCRIPTION:
Medical advances in the treatment of HIV/AIDS have improved the life expectancy of HIV-infected individuals. Unfortunately, HIV-infected individuals are three times more likely to use tobacco than those in the general population, but little is known about the mechanisms that underlie these high smoking rates. This will be the first study to test whether the neurocognitive impairments associated with HIV-1 infection may be exacerbated during nicotine withdrawal and increase the probability of smoking relapse among HIV-infected smokers (HIV+), compared to HIV-uninfected smokers (HIV-). To this end, adult treatment-seeking smokers (N=300; 150 HIV+ and 150 HIV-) will complete this 12-week study, which is divided into two phases: a pre-quit laboratory phase (weeks 0-2) and a treatment phase (weeks 3-12). Subjects will complete two laboratory sessions during the pre-quit phase: once following 24 hours of mandatory smoking abstinence and once while smoking-as-usual (order counterbalanced). A comprehensive cognitive task battery assessing memory, attention, and executive function will be administered during each laboratory session. During the treatment phase, all subjects will receive standard smoking cessation treatment, including counseling (weeks 3-8) and open-label transdermal nicotine (TN) patches (weeks 4-12). The primary outcomes are: 1) cognitive performance following 24-hours smoking abstinence (vs. smoking-as-usual) during the pre-quit phase; and 2) 7-day point-prevalence, biochemically-confirmed abstinence rates at the end-of-treatment (EOT) for the treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or older who self-report smoking at least 5 cigarettes (menthol and non-menthol) per day, on average.
* HIV status

  1. HIV-infected smokers: diagnosed with HIV infection and exhibiting viral load of less than or equal to 1000 copies/mL and CD4+ counts of greater than or equal to 200 cells/mm3 within 12 months prior to enrollment.
  2. HIV-uninfected smokers: negative HIV status will be confirmed by an on-site rapid HIV blood test.
* Able to use transdermal nicotine (TN) safely, based on a medical evaluation.
* Residing in the geographic area for at least 4 months.
* Women of childbearing potential (based on medical history) must consent to use a medically accepted method of birth control (e.g., condoms and spermicide, oral contraceptive, Depo-Provera injection, contraceptive patch, tubal ligation) or abstain from sexual intercourse during the time they are in the study and using transdermal nicotine.
* Able to communicate fluently in English.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent/HIPAA form.

Exclusion Criteria:

Smoking Behavior

1. Current enrollment or plans to enroll in another smoking cessation program in the next 4 months.
2. Regular (daily) use of electronic cigarettes, chewing tobacco, snuff, snus, cigars, cigarillos, or pipes.
3. Current use or plans to use nicotine substitutes (gum, patch, lozenge, e-cigarette) or smoking cessation treatments in the next 4 months.

Alcohol/Drug Exclusion Criteria

1. Current untreated and unstable diagnosis of substance dependence (eligible if past use and if receiving treatment and stable for at least 30 days). Current untreated and unstable diagnosis of substance abuse requires Study Physician approval.
2. A positive urine drug screen for cocaine, amphetamines, methamphetamines, Phencyclidine (PCP), barbiturates, ecstasy (MDMA) at Intake (see Measures and Table 1 for details). At Lab 1 and Lab 2, positive urine drug screens will be reviewed on a case-by-case basis. The PI will determine if the participant will be excluded or allowed to reschedule the visit, at which time they must provide a negative drug screen to continue with the study.

Medication Exclusion Criteria

Current use or recent discontinuation (within last 14 days) of the following medications:

1. Other smoking cessation medications (e.g. Zyban, Wellbutrin, Wellbutrin sustained release (SR), Chantix)

   a. Note: Once participants are found eligible for the study, they are instructed to only use the NRT provided to them by the study staff. If a subject reports using a non-study smoking cessation medication (including other forms of NRT), the study physician and PI will evaluate the situation and determine if it is safe for the subject to continue participation.
2. Anti-psychotic medications (if used to treat psychotic symptoms. Other uses may be eligible pending physician approval).
3. Daily use of opiate-containing medications for chronic pain (Duragesic/fentanyl patches, Percocet, Oxycontin). Smokers who report taking opiate-containing medications on an "as-needed" basis will be instructed to refrain from use until their study participation is over and that they will be tested to ensure they have complied with this requirement.
4. Asthma medications/corticosteroids (requires physician approval)
5. Anti-depressants (require physician approval)

Medical Exclusion Criteria

1. Females who self-report current pregnancy, planning a pregnancy during the study, or currently breastfeeding/lactating.
2. Current diagnosis of unstable and untreated major depression, as determined by self-report & Mini International Neuropsychiatric Interview (MINI) (eligible if stable for at least 30 days).
3. Current or past diagnosis of bipolar disorder or psychotic disorder, as determined by self-report or MINI.
4. History of heart disease, stroke or MI, unstable angina, or tachycardia (if stable, requires Study Physician approval).
5. Uncontrolled hypertension (systolic blood pressure (SBP) greater than 160 or diastolic blood pressure (DBP) greater than 100) present at Intake.

   a. Note: If a participant presents with blood pressure greater than 160/100 at sessions occurring on Week 3 (Pre-Quit) or at any other point during the treatment period, they will not be provided with/able to continue on TN unless the study physician grants approval.
6. Previous allergic reaction to TN.
7. History of diabetes (requires Study Physician approval)
8. History of seizures (requires Study Physician approval)
9. History of stomach ulcers (requires Study Physician approval)

Suicide History Exclusion Criteria

1. Suicide risk as indicated by at least one of the following on the Columbia Suicide Severity Rating Scale (the PI &/or study psychologist will be consulted to assess safety and determine eligibility in cases close to the eligibility cutoffs):

1. Current suicidal ideation (within 30 days of enrollment)
2. Two or more lifetime suicide attempts
3. Any suicide attempt within 2 years of enrollment

General Exclusion Criteria

1. Any medical condition or concomitant medication that could compromise subject safety or treatment, as determined by the Principal Investigator and/or Study Physician.
2. Color blindness.
3. Any impairment (physical and/or neurological) including visual or other impairment preventing cognitive task performance.
4. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator and/or Study Physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three hundred (150 HIV+ and 150 HIV-) adult male and female smokers 18 years of age or older who smoke at least 5 cigarettes per day and are interested in quitting smoking will complete the study. HIV-infected smokers have been diagnosed with HIV/AIDS and HIV-uninfected smokers will have no diagnosis of HIV, either via blood test or self-report.
Sampling Method: Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Ashare, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greene B, Schnoll RA, Gross R, Ashare RL. The role of alternative reinforcers in smoking outcomes among people with and without HIV. Psychol Addict Behav. 2025 Nov;39(7):632-643. doi: 10.1037/adb0001071. Epub 2025 Jun 5. PMID 40471817

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV+, Smoking Lab Session First, Abstinence Lab Session Second, Then Treatment: HIV-infected smokers: diagnosed with HIV infection and exhibiting viral load of less than or equal to 1000 copies/mL and CD4+ counts of greater than or equal to 200 cells/mm3 within 6 months prior to enrollment
  Participants were randomized to complete a smoking-as-usual lab session first followed by a 24-hour abstinence lab session second. All participants then received treatment.
  Treatment:
  Nicotine patch: All participants will receive nicotine patches to aid in quitting smoking. TN is available over the counter and is very well tolerated. Participants will use "the patch" in a tapering fashion as recommended by the manufacturer. Participants who smoke 10 or more cigarettes per day will adhere to the following dosing guidelines: 21 mg for 4 weeks; 14 mg for 2 weeks and 7 mg for 2 weeks. Individuals who smoke between 5 and 9 cigarettes per day will follow a modified dosing regimen: 14 mg for 6 weeks and 7 mg for 2 weeks.
  Behavioral counseling: Participants will attend 6 counseling sessions and receive standard smoking cessation counseling (SC).
- HIV-, Smoking Lab Session First, Abstinence Lab Session Second, Then Treatment: HIV-uninfected smokers: negative HIV status will be confirmed by an on-site rapid HIV blood test
  Participants were randomized to complete a smoking-as-usual lab session first followed by a 24-hour abstinence lab session second. All participants then received treatment.
  Treatment:
  Nicotine patch: All participants will receive nicotine patches to aid in quitting smoking. TN is available over the counter and is very well tolerated. Participants will use "the patch" in a tapering fashion as recommended by the manufacturer. Participants who smoke 10 or more cigarettes per day will adhere to the following dosing guidelines: 21 mg for 4 weeks; 14 mg for 2 weeks and 7 mg for 2 weeks. Individuals who smoke between 5 and 9 cigarettes per day will follow a modified dosing regimen: 14 mg for 6 weeks and 7 mg for 2 weeks.
  Behavioral counseling: Participants will attend 6 counseling sessions and receive standard smoking cessation counseling (SC).
- HIV+, Abstinence Lab Session First, Smoking-as-usual Second, Then Treatment: HIV-infected smokers: diagnosed with HIV infection and exhibiting viral load of less than or equal to 1000 copies/mL and CD4+ counts of greater than or equal to 200 cells/mm3 within 6 months prior to enrollment
  Participants were randomized to complete a 24-hour abstinence lab session first, followed by a smoking-as-usual lab session second. All participants then received treatment.
  Treatment:
  Nicotine patch: All participants will receive nicotine patches to aid in quitting smoking. TN is available over the counter and is very well tolerated. Participants will use "the patch" in a tapering fashion as recommended by the manufacturer. Participants who smoke 10 or more cigarettes per day will adhere to the following dosing guidelines: 21 mg for 4 weeks; 14 mg for 2 weeks and 7 mg for 2 weeks. Individuals who smoke between 5 and 9 cigarettes per day will follow a modified dosing regimen: 14 mg for 6 weeks and 7 mg for 2 weeks.
  Behavioral counseling: Participants will attend 6 counseling sessions and receive standard smoking cessation counseling (SC).
- HIV-, Abstinence Lab Session First, Smoking-as-usual Second, Then Treatment: HIV-uninfected smokers: negative HIV status will be confirmed by an on-site rapid HIV blood test
  Participants were randomized to complete a 24-hour abstinence lab session first, followed by a smoking-as-usual lab session second. All participants then received treatment.
  Treatment:
  Nicotine patch: All participants will receive nicotine patches to aid in quitting smoking. TN is available over the counter and is very well tolerated. Participants will use "the patch" in a tapering fashion as recommended by the manufacturer. Participants who smoke 10 or more cigarettes per day will adhere to the following dosing guidelines: 21 mg for 4 weeks; 14 mg for 2 weeks and 7 mg for 2 weeks. Individuals who smoke between 5 and 9 cigarettes per day will follow a modified dosing regimen: 14 mg for 6 weeks and 7 mg for 2 weeks.
  Behavioral counseling: Participants will attend 6 counseling sessions and receive standard smoking cessation counseling (SC).
Period: Lab Session 1 (Week 1)
Arm/Group | HIV+, Smoking Lab Session First, Abstinence Lab Session Second, Then Treatment | HIV-, Smoking Lab Session First, Abstinence Lab Session Second, Then Treatment | HIV+, Abstinence Lab Session First, Smoking-as-usual Second, Then Treatment | HIV-, Abstinence Lab Session First, Smoking-as-usual Second, Then Treatment
Started | 41 | 77 | 43 | 80
Completed | 41 | 77 | 43 | 76
Not Completed | 0 | 0 | 0 | 4
Not completed — Protocol Violation | 0 | 0 | 0 | 4
Period: Lab Session 2 (Week 2)
Arm/Group | HIV+, Smoking Lab Session First, Abstinence Lab Session Second, Then Treatment | HIV-, Smoking Lab Session First, Abstinence Lab Session Second, Then Treatment | HIV+, Abstinence Lab Session First, Smoking-as-usual Second, Then Treatment | HIV-, Abstinence Lab Session First, Smoking-as-usual Second, Then Treatment
Started | 41 | 77 | 43 | 76
Completed | 39 | 60 | 41 | 70
Not Completed | 2 | 17 | 2 | 6
Period: Treatment Phase (Weeks 3-12)
Arm/Group | HIV+, Smoking Lab Session First, Abstinence Lab Session Second, Then Treatment | HIV-, Smoking Lab Session First, Abstinence Lab Session Second, Then Treatment | HIV+, Abstinence Lab Session First, Smoking-as-usual Second, Then Treatment | HIV-, Abstinence Lab Session First, Smoking-as-usual Second, Then Treatment
Started | 39 | 59 (One participant was lost to follow-up between the end of the laboratory phase and the start of the treatment phase) | 41 | 68 (Two participants were lost to follow-up between the end of the laboratory phase and the start of the treatment phase)
Completed | 38 | 48 | 37 | 63
Not Completed | 1 | 11 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- HIV+: HIV-infected smokers: diagnosed with HIV infection and exhibiting viral load of less than or equal to 1000 copies/mL and CD4+ counts of greater than or equal to 200 cells/mm3 within 6 months prior to enrollment
  Nicotine patch: All participants will receive nicotine patches to aid in quitting smoking. TN is available over the counter and is very well tolerated. Participants will use "the patch" in a tapering fashion as recommended by the manufacturer. Participants who smoke 10 or more cigarettes per day will adhere to the following dosing guidelines: 21 mg for 4 weeks; 14 mg for 2 weeks and 7 mg for 2 weeks. Individuals who smoke between 5 and 9 cigarettes per day will follow a modified dosing regimen: 14 mg for 6 weeks and 7 mg for 2 weeks.
  Behavioral counseling: Participants will attend 6 counseling sessions and receive standard smoking cessation counseling (SC).
- HIV-: HIV-uninfected smokers: negative HIV status will be confirmed by an on-site rapid HIV blood test
  Nicotine patch: All participants will receive nicotine patches to aid in quitting smoking. TN is available over the counter and is very well tolerated. Participants will use "the patch" in a tapering fashion as recommended by the manufacturer. Participants who smoke 10 or more cigarettes per day will adhere to the following dosing guidelines: 21 mg for 4 weeks; 14 mg for 2 weeks and 7 mg for 2 weeks. Individuals who smoke between 5 and 9 cigarettes per day will follow a modified dosing regimen: 14 mg for 6 weeks and 7 mg for 2 weeks.
  Behavioral counseling: Participants will attend 6 counseling sessions and receive standard smoking cessation counseling (SC).
- Total: Total of all reporting groups
Arm/Group | HIV+ | HIV- | Total
Number analyzed (Participants) | 93 | 181 | 274
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 88 | 166 | 254
  >=65 years | 5 | 15 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (9.4) | 51.6 (11.4) | 51.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 80 | 109
  Male | 64 | 101 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 87 | 174 | 261
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 84 | 125 | 209
  White | 3 | 39 | 42
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 3 | 12 | 15
Region of Enrollment [Number; unit: participants]
  United States | 93 | 181 | 274
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 11.6 (5.4) | 13.3 (6.2) | 12.7 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Function
Description: Cognitive function will be assessed at the Lab session 1 and lab session 2 visits as well as End of Treatment. Participants will complete measures of executive function, verbal learning and memory and response inhibition. The primary outcome is the change in cognitive function lab session 1, lab session 2, and End of Treatment measured by a composite score (calculated by averaging individual z-scores). Z-scores were calculated using the Stroop interference score (executive function; measured in milliseconds), the delayed recall score from the Hopkins Verbal Learning Test (verbal learning and memory), and the Stop signal reaction time from the Stop Signal Task (response inhibition, measured in milliseconds). A composite score will be created by computed standardized z-scores for each measure (where the mean is 0 and the standard deviation is 1) and then averaging the z-scores. Measures of response time were reverse coded such that higher z-scores indicate better cognitive performance.
Time Frame: Lab session 1 (week 1), lab session 2 (week 2), End of treatment (week 12)
Population: Numbers are different due to attrition between enrollment and lab session 1. Some cognitive data were excluded due to outliers.
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- HIV+ Smoking Lab Session First: HIV-infected smokers: diagnosed with HIV infection and exhibiting viral load of less than or equal to 1000 copies/mL and CD4+ counts of greater than or equal to 200 cells/mm3 within 6 months prior to enrollment
  Randomized to complete smoking-as-usual lab session first and 24-h abstinent lab session second
  Nicotine patch: All participants will receive nicotine patches to aid in quitting smoking. TN is available over the counter and is very well tolerated. Participants will use "the patch" in a tapering fashion as recommended by the manufacturer. Participants who smoke 10 or more cigarettes per day will adhere to the following dosing guidelines: 21 mg for 4 weeks; 14 mg for 2 weeks and 7 mg for 2 weeks. Individuals who smoke between 5 and 9 cigarettes per day will follow a modified dosing regimen: 14 mg for 6 weeks and 7 mg for 2 weeks.
  Behavioral counseling: Participants will attend 6 counseling sessions and receive standard smoking cessation counseling (SC).
- HIV- Smoking Lab Session First: HIV-uninfected smokers: negative HIV status will be confirmed by an on-site rapid HIV blood test
  Randomized to complete smoking-as-usual lab session first and 24-h abstinent lab session second
  Nicotine patch: All participants will receive nicotine patches to aid in quitting smoking. TN is available over the counter and is very well tolerated. Participants will use "the patch" in a tapering fashion as recommended by the manufacturer. Participants who smoke 10 or more cigarettes per day will adhere to the following dosing guidelines: 21 mg for 4 weeks; 14 mg for 2 weeks and 7 mg for 2 weeks. Individuals who smoke between 5 and 9 cigarettes per day will follow a modified dosing regimen: 14 mg for 6 weeks and 7 mg for 2 weeks.
  Behavioral counseling: Participants will attend 6 counseling sessions and receive standard smoking cessation counseling (SC).
- HIV+ Abstinent Lab Session First: Same as HIV+ Smoking lab session first except Randomized to complete 24-h abstinent lab session first and smoking-as-usual lab session second
- HIV- Abstinent Lab Session First: Same as HIV- Smoking lab session first except Randomized to complete 24-h abstinent lab session first and smoking-as-usual lab session second
Arm/Group | HIV+ Smoking Lab Session First | HIV- Smoking Lab Session First | HIV+ Abstinent Lab Session First | HIV- Abstinent Lab Session First
Number analyzed (Participants) | 41 | 77 | 43 | 75
z-score
  Lab session 1 (week 1) | 0.125 (0.489) | -.093 (0.441) | -.059 (.452) | -.008 (.553)
  Lab session 2 (week 2): number analyzed (Participants) | 39 | 60 | 41 | 70
  Lab session 2 (week 2) | .043 (.498) | -.012 (.441) | -.106 (.488) | .014 (.546)
  End of treatment (week 12): number analyzed (Participants) | 37 | 42 | 36 | 59
  End of treatment (week 12) | 0.149 (.416) | -.082 (.465) | -.091 (.440) | .001 (.559)

2. Secondary Outcome: 7-day Point Prevalence Abstinence
Description: Smoking abstinence (primary outcome) will be assessed and biochemically verified at the End of Treatment Visit (week 12). The primary smoking outcome variable will be 7-day point prevalence abstinence (no smoking, not even a puff, for at least 7 days prior to the assessment) biochemically verified by carbon monoxide < 5 ppm.
Time Frame: End of Treatment (week 12)
Population: Only subjects who entered treatment following the two lab sessions were considered intent to treat and included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+ | HIV-
Number analyzed (Participants) | 80 | 127
Participants | 22 | 33

ADVERSE EVENTS:
Time Frame: 12 weeks: From the start of treatment through end of treatment
Description: Adverse event reporting was completed using a symptom checklist, listing all expected side effects for the study drug. It was administered once treatment was initiated after both lab sessions were completed. Participants were also given an open-ended item. Groups do not distinguish by "lab session order" because the lab sessions were completed prior to the initiation of any treatment, so they are combined into HIV+ and HIV- only.
Arm/Group | HIV+ | HIV-
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/127
Serious Adverse Events (participants affected / at risk) | 0/80 | 2/127
Other Adverse Events (participants affected / at risk) | 32/80 | 36/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV+ (N=80) | HIV- (N=127)
Stroke (Cardiac disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV+ (N=80) | HIV- (N=127)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 10 (24) | 6 (31)
Itching, burning or tingling at patch site (Skin and subcutaneous tissue disorders) | 6 (12) | 7 (8)
Skin redness (Skin and subcutaneous tissue disorders) | 9 (16) | 2 (3)
Sleep disturbances (General disorders) | 13 (32) | 24 (48)
Vivid dreams (General disorders) | 9 (13) | 13 (25)
Weakness (General disorders) | 6 (7) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT03169101/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT03169101/ICF_001.pdf